CLINICAL TRIAL: NCT06982911
Title: Comparison of Postoperative Pulmonary Complications Between Smokers and Nonsmokers: A Prospective Cohort Study
Brief Title: Comparison of Postoperative Pulmonary Complications Between Smokers and Nonsmokers
Acronym: MINOPPC
Status: Completed | Type: Observational
Sponsor: mehmet özkılıç (Other)
Responsible Party: Sponsor-Investigator, mehmet özkılıç, Specialist in Anesthesiology and Reanimation, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Organization: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Other Study IDs: GYEAH-PPC-001
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Coughing; Post Operative Complications; Wheezing; Smoking, Tobacco
Keywords: Smoking; Pulmonary Secretions; Postoperative Complication; Cough; Abdominal Surgery
MeSH Terms: conditions — Cough; Respiratory Sounds; Tobacco Smoking; Smoking; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smoking Group: Patients with an active smoking history (defined as smoking ≥10 pack-years) undergoing elective abdominal surgery under general anesthesia. This group will be evaluated for early postoperative respiratory symptoms such as increased secretions, cough, and wheezing.
- Nonsmoking Group: Patients with no active smoking history (never smoked or quit more than 1 year ago) undergoing elective abdominal surgery under general anesthesia. This group serves as the control and will be assessed using the same early postoperative respiratory criteria.

SUMMARY:
This is a prospective observational study designed to evaluate the effect of smoking on early postoperative respiratory symptoms such as cough, airway secretions, and wheezing in adult patients undergoing elective abdominal surgery. Participants will be divided into two groups based on smoking history. The study aims to assess the incidence of minor pulmonary complications-such as increased secretions requiring suctioning, oxygen need, and early respiratory discomfort-within the first 24 hours after surgery. Data will be collected on parameters including secretion volume, oxygen saturation, aspiration frequency, and presence of cough or wheezing. The results will help determine whether active smoking is associated with a higher frequency of early postoperative pulmonary events.

DETAILED DESCRIPTION:
Cigarette smoking is a well-established risk factor for adverse postoperative outcomes, including respiratory complications. However, many studies have primarily focused on major complications such as pneumonia, reintubation, or prolonged mechanical ventilation, often underestimating early and subtle pulmonary effects of smoking. This study aims to fill that gap by evaluating early minor postoperative pulmonary events-specifically cough, airway secretions, and wheezing-within the first 24 hours after extubation in adult patients undergoing elective abdominal surgery.

The study is designed as a prospective observational cohort conducted in a single tertiary-care hospital. Adult patients (aged 18-65) undergoing elective abdominal surgery under general anesthesia will be included. Participants will be classified into two groups based on smoking history: current smokers and non-smokers. The primary outcome is the occurrence of early minor pulmonary complications, including secretion burden requiring aspiration, Peripheral Oxygen Saturation(SpO₂ ) desaturation (SpO₂ <90%), presence of audible wheezing, and persistent postoperative cough. These events will be documented by trained clinical staff using standardized clinical criteria and data collection forms.

The hypothesis of this study is that active smokers are more likely to develop early minor pulmonary complications within the first 24 hours after surgery compared to non-smokers. The findings will contribute to a better understanding of early perioperative respiratory risk among smoking patients and may support the refinement of risk assessment and preoperative counseling.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Undergoing elective abdominal surgery under general anesthesia
* ASA physical status I-II-III
* Able to provide informed consent
* Classified as either active smoker (≥10 pack-years) or nonsmoker (never smoked or quit >1 year ago)

Exclusion Criteria:

* Diagnosed chronic pulmonary disease (e.g., Obstructive Sleep Apnea, asthma, Chronic Obstructive Pulmonary Disease)
* Acute respiratory tract infection within the past 30 days
* Morbid obesity (Body Mass Index >35 kg/m²)
* Emergency surgery
* Pregnancy or breastfeeding
* Refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients between 18 and 60 years old scheduled for elective abdominal surgery at a tertiary care hospital. Participants include both current smokers and nonsmokers. All patients are American Society of Anesthesiologists (ASA) class I-II-III and free of known chronic respiratory diseases.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Early Postoperative Pulmonary Complications Within 24 Hours After Surgery | Within the first 24 hours after extubation
  The primary outcome is defined as the presence of at least one of the following respiratory findings within 24 hours after extubation: (1) increased airway secretions requiring aspiration, (2) persistent cough, (3) audible wheezing, or (4) oxygen desaturation below 90% on room air. These events will be documented by trained clinical staff using a standardized data collection form. Each patient will be assessed continuously for the first 6 hours and again at the 24th postoperative hour. The incidence of these pulmonary complications will be compared between smoking and nonsmoking patients.

SECONDARY OUTCOMES:
Number of Suctions Required for Airway Secretion Clearance Within 6 Hours After Extubation | Within the first 1 hours after extubation
  This outcome measures the total number of suctioning procedures required to clear airway secretions during the first 6 hours after extubation. Suctioning is performed only when visible or audible secretions are present and is recorded by trained clinical staff using a standardized protocol.
Oxygen Desaturation Events Below 90% Within the First 24 Hours After Surgery | Within the first 24 hours after extubation
  This outcome tracks the number and duration of oxygen desaturation episodes defined as saturation(SpO₂) falling below 90% on room air within the first 24 hours after extubation. Each event is recorded by trained clinical personnel using pulse oximetry. Desaturation episodes that are corrected by airway maneuvers or supplemental oxygen are noted.
Association Between Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) Risk Score and Postoperative Pulmonary Complications | Within the first 24 hours after surgery
  The Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) score will be calculated preoperatively for all included patients using seven validated clinical parameters (age, preoperative saturation (SpO2), respiratory infection in the last month, preoperative anemia, surgical incision type, duration of surgery, and emergency status). This score will be evaluated as a secondary outcome to assess its correlation with the incidence of early postoperative pulmonary complications (PPCs). The score will also be included in multivariate analysis models and ROC curve analysis to determine predictive value and optimal cutoff thresholds.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi Yaşargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this is a single-center, observational study and no explicit consent for data sharing was obtained from participants. Only aggregate results will be published.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT06982911/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT06982911/ICF_001.pdf